CLINICAL TRIAL: NCT05947669
Title: Efficacy and Safety of Infliximab for Immune Checkpoint Inhibitor Induced Colitis: a Multinational, Randomised, Open Label, Phase III Trial - The iCaD Study
Brief Title: Efficacy and Safety of Infliximab for Immune Checkpoint Inhibitor Induced Colitis
Acronym: iCaD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The ICaD Study
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Colitis
MeSH Terms: conditions — Colitis | interventions — Infliximab; Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care - Methylprednisolone (Active Comparator): Subjects are hospitalised Day 1 and for at least 4 days. It is accepted that participating centres handle the subjects on an outpatient basis as long as all study requirements are met. Methylprednisolone 80 mg intravenously (body weight 40-80 kg; methylprednisolone 1 mg/kg if body weight < 40 or > 80 kg) will be administered from Day 1 until mCTCAE ir-colitis/diarrhoea grade ≤ 2 and hereafter converted to oral prednisolone. During tapering, if ir-colitis/diarrhoea increases from grade 2 to ≥ grade 3, or from grade < 2 to ≥ grade 2, re-assessment including diagnostic workup will be performed, and the patient will be evaluated for rescue infliximab.
  Interventions: Drug: Methylprednisolone; Drug: Prednisolone
- Treatment with infliximab (Experimental): Infliximab will be administered Day 1 or latest Day 2 (within 48 hours). Infliximab infusion is handled as standard by skilled staff. A second dose of infliximab will be administered if ir-colitis/diarrhoea has not resolved to grade ≤ 2 on Day 7. Methylprednisolone 80 mg (body weight 40-80 kg; methylprednisolone 1 mg/kg if body weight < 40 or > 80 kg) intravenously is co-administered from Day 1 until mCTCAE ir-colitis/diarrhoea grade ≤ 2 and hereafter converted to oral prednisolone. Initial dosage of infliximab is 5 mg/kg. Dosage of infliximab for subjects referred to a second dose of infliximab will be left to the discretion of the treating physician. In the event of failure of infliximab, second line biological immunosuppressant treatment will also be left to the discretion of the treating physician.
  Interventions: Drug: Infliximab; Drug: Methylprednisolone; Drug: Prednisolone

INTERVENTIONS:
Drug: Infliximab — Infliximab is available in vials of 100 mg with pharmaceutical form of concentrate for solution for infusion. Participating sites will ensure availability of infliximab as part of the hospital's standard supply for use in the study.
  Arms: Treatment with infliximab
Drug: Methylprednisolone — Methylprednisolone is available in vials of 40 mg. Methylprednisolone is a drug used for standard treatment first line for ir-colitis or diarrhoea CTCAE grade ≥ 3. Participating sites will ensure availability of methylprednisolone for use in the study as part of the hospitals standard supply.
Drug: Prednisolone — Prednisolone is available in tablets of 25 or 5 mg. Oral corticosteroids are internationally recommended as initial treatment for ir-colitis and ir-diarrhoea CTCAE grade 2 [24-27]. Participating sites will ensure availability of prednisolone for use in the study as part of the hospitals' standard supply.

SUMMARY:
The goal of this clinical trial is to assess whether the early introduction of biological treatment with a TNF-alpha inhibitor (infliximab) in addition to corticosteroids for severe ir-colitis/diarrhoea will reduce the time to grade ≤ 1 ir-colitis/diarrhoea compared to corticosteroids alone in patients scheduled for ICI treatment for solid tumors and untreated mCTCAE grade 2-4 diarrhoea or colitis.

The main question it aims to answer is:

• Can an early introduction of biological treatment with a TNF-alpha inhibitor (infliximab) in addition to corticosteroids reduce the time to grade ≤ 1 ir-colitis/diarrhoea compared to corticosteroids alone.

Participants will be randomised 1:1:

Arm A: All patients will receive same dose of methylprednisolone i.v. daily. Arm B: Patients allocated to Arm B will in addition receive infliximab i.v. day 1 or 2.

Study patients are evaluated with blood samples, faecal samples and by sigmoidoscopy. Procedures are performed before randomisation and as part of follow up.

ELIGIBILITY:
Inclusion Criteria

* Untreated mCTCAE grade 2-4 diarrhoea or colitis, or persistent mCTCAE grade 2 diarrhoea after administration of loperamide or equivalent for mCTCAE grade ≤ 2 diarrhoea
* No signs of colonic perforation or infection
* Age ≥ 18
* Understands the nature and purpose of the study and the study procedures and has signed informed consent
* Is able to read, understand, and complete questionnaires and daily components of the patient Diary for the study period
* Histologically confirmed malignant solid tumours
* Treatment with immune checkpoint inhibitors (anti-CTLA-4, anti-PD-1 or anti-PD-L1) within the past 12 weeks. Immune checkpoint inhibitors can be administered as single agents or as combination therapy with anti-CTLA-4 and anti-PD-1
* No probability of a concomitant treatment (e.g. laxatives) other than the immune checkpoint inhibitor being the causal drug for the colitis or diarrhoea
* Prior treatment with immune checkpoint inhibitors is allowed
* Usage of prednisolone ≤ 10 mg daily for non irAE is allowed
* Diagnostic work up including screening for viral hepatic infection and QuantiFERON-TB for mycobacterium tuberculosis must be requisitioned but will not need to be reported prior to study enrolment
* Women of child bearing potential must have a negative serum (preferred) or urine pregnancy test within 72 hours prior to registration.

  * Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and after the study treatment:

  * for at least 6 months after the last study treatment, or depending on the duration antineoplastic treatment
  * Note: A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Sexual abstinence

Exclusion Criteria

* Prior history of inflammatory bowel disease, colitis, or diarrhoea requiring treatment with any corticosteroid, or any other immunosuppressant medication
* Prior history of recurrent bowel disease including symptomatic diverticulosis
* Current positive testing for Clostridium difficile or other colonic infection
* Current bacterial infection requiring antibiotic treatment, or systemic fungal infection
* Ongoing antibiotic treatment for any reason
* Treatment with systemic corticosteroids within the last four weeks prior to study enrolment (daily usage of prednisolone ≤ 10 mg for non irAE conditions is accepted)
* Concurrent immune-related adverse events requiring immunosuppressant medication of any kind
* Known hypersensitivity or contraindications to systemic corticosteroids or infliximab
* Prior history of viral hepatitis with a positive viral load, known untreated mycobacterium tuberculosis, or known active herpes zoster infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Time (days) to persistent modified CTCAE grade ≤ 1 ir-colitis/diarrhoea. | From the first day of grade ≤ 1 ir-colitis/diarrhoea of that period (time frame: seven weeks)
  Persistent is defined as grade ≤ 1 ir-colitis/diarrhoea for five consecutive days or more with no increase in corticosteroid intake

SECONDARY OUTCOMES:
Proportion of study subjects with grade ≤ 1 ir-colitis/diarrhoea at 72 hours. | Time frame: 72 hours
Proportion of study subjects with persistent grade ≤ 1 ir-colitis/diarrhoea at three weeks. | The event will be calculated from the first day of grade ≤ 1 ir-colitis/diarrhoea of that period (time frame: three weeks)
  Persistent is defined as grade ≤ 1 ir-colitis/diarrhoea for five consecutive days or more
Proportion of study subjects with a corticosteroid-free clinical remission (grade ≤ 1 ir-colitis/diarrhoea) after seven weeks. | Time frame: seven weeks
Proportion of study subjects requiring rescue immunosuppressive medication | Time frame: seven days
  Arm A (initial corticosteroid only): infliximab if no improvement to grade ≤ 2 ir-colitis/diarrhoea after 3 days (time frame: seven weeks); Arm B (initial infliximab): second dose infliximab according to physicians decision if no improvement to grade ≤ 2 ir-colitis/diarrhoea after seven days
Cumulative corticosteroid exposure | Time frame: seven weeks
QoL by means of EORTC-QLQ-C30 | Change in score from baseline to 3, 12, 24, and 52 weeks after randomisation
  A 30-item questionaire developed to assess the quality of life of cancer patients. Item 1-28 is scaled in a 4 scale score from 'not at all' to 'very much'. Item 29-30 is a numeric rating scale from 1 to 7 assessing overall health/quality of life. One denotes very poor and 7 denotes excellent.
  Measure: changes in quality of life
QoL by means of selected PRO-CTCAE items | Change in score from baseline to 3, 12, 24, and 52 weeks after randomisation
  A 8 item questionnaire assessing bowel related issues. The scales ranges from eg:
  Yes/No Never/rarely/occasionally/frequently/almost constant None/mild/moderate/severe/very severe Not at all/a little bit/ somewhat/quit a bit/very much Measure: changes in bowel related symptoms
Proportion of study subjects with treatment related adverse events as assessed by CTCAE v5.0 | Time frame: 12 weeks
Proportion of study subjects with colectomy or colitis-specific mortality | Time frame: seven weeks

OTHER OUTCOMES:
Proportion of study subjects with recurrence of ir-colitis/diarrhoea on subsequent reintroduction of ICI. | Timeframe: Up to 24 weeks
Subgroup analyses stratified for ipilimumab containing ICI for time (days) to persistent grade ≤ 1 ir-colitis/diarrhoea. | week 3
  Persistent is defined as grade ≤ 1 ir-colitis/diarrhoea for five consecutive days or more.
Progression Free Survival stratified by cancer type | Time frame: duration of time from start of randomisation to time of progression or death, whichever occurs first or up to 24 months
Overall Survival stratified by cancer type | Time frame: the duration of time from start of randomisation to time of death or up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina H. Ruhlmann, PhD, Principal Investigator — Department of Oncology, OUH
Locations (3):
- Denmark (2):
  - Department of Oncology, Aalborg University Hospital, Aalborg
  - Department of Oncology Odense University Hospital, Odense
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Prior to study initiation, the study will be registered at www.clinicaltrials.gov. No later than six months after Follow-up completion, a study report will be completed and data displayed on www.clinicaltrials.gov. Study results will be submitted to the Clinical Trials Information System (CTIS) portal as soon as possible and no later than one year after the trial has ended. In addition, the anonymised data will be made public available through the Zenodo open data repository (CERN), or an equivalent public database.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: No later than one year after the trial has ended.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT05947669/Prot_SAP_000.pdf